CLINICAL TRIAL: NCT05044962
Title: Co-benefits of Co-delivery of Long-acting Antiretrovirals and Contraceptives
Brief Title: Kuwa Free! - Live Free!
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Moi Teaching and Referral Hospital (Other); Indiana University (Other); University of Nebraska (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Rena Patel, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00012640; R01AI155052 (NIH)
Record Dates: First submitted 2021-08-26; First posted 2021-09-16 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: HIV Infections; Contraception; Drug-drug Interaction
Keywords: Kenya; Adolescent girls and young women; HIV adherence; Long-acting antiretroviral therapy; Injectable cabotegravir; Injectable rilpivirine
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir; Rilpivirine; etonogestrel; Levonorgestrel

STUDY DESIGN:
Intervention Model Description: The hybrid trial will be a parallel, randomized design.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and care providers will not be masked (open label), but the principle and site-principal investigators and study statistician will be blinded to arm allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Aim 1a (PK study group 1) (Experimental): Initiating injectable cabotegravir/rilpivirine (LA ART) and DMPA
  Interventions: Drug: Cabotegravir/ Rilpivirine; Drug: Intramuscular depo-medroxyprogesterone acetate (IM DMPA)
- Aim 1a (PK study group 2) (Experimental): Initiating injectable cabotegravir/rilpivirine (LA ART) and and etonogestrel implant
  Interventions: Drug: Cabotegravir/ Rilpivirine; Drug: Etonogestrel (ETG) implant
- Aim 1a (PK study group 3) (Experimental): Initiating injectable cabotegravir/rilpivirine (LA ART) and levonorgestrel implant.
  Interventions: Drug: Cabotegravir/ Rilpivirine; Drug: Levonorgestrel
- Aim 1a (PK study group 4) (Active Comparator): Receiving injectable cabotegravir/ rilpivirine (LA ART) and not using any hormonal contraceptive method (e.g. copper IUD)
  Interventions: Drug: Cabotegravir/ Rilpivirine
- Aim 1a (PK study group 5) (Active Comparator): AGYW without HIV and not exposed to antiretrovirals (e.g., for PrEP) initiating DMPA
  Interventions: Drug: Intramuscular depo-medroxyprogesterone acetate (IM DMPA)
- Aim 2a (Hybrid trial intervention group) (Experimental): AGYW with viral suppression on their current ART regimen to switch to cabotegravir/ rilpivirine.
  Interventions: Drug: Cabotegravir/ Rilpivirine
- Aim 2a (Hybrid trial comparator group) (Active Comparator): AGYW with viral suppression to continue their oral ART regimen.
  Interventions: Drug: NNRTI, PI, or INSTI-containing 1st or 2nd line ART regimens

INTERVENTIONS:
Drug: Cabotegravir/ Rilpivirine — For initial injection participants will be given CABENUVA 600-mg/900-mg Kit: (single-dose vial of 600 mg/3 mL (200 mg/mL) cabotegravir , single-dose vial of 900 mg/3 mL (300 mg/mL) rilpivirin).
  For subsequent injections participants will be given CABENUVA 400-mg/600-mg Kit: (single-dose vial of 400 mg/2 mL (200 mg/mL) cabotegravir, single-dose vial of 600 mg/2 mL (300 mg/mL) rilpivirine)
  CABENUVA® is owned by or licensed to the ViiV Healthcare group of companies, GlaxoSmithKline Research Triangle Park, NC 27709
  Arms: Aim 1a (PK study group 1); Aim 1a (PK study group 2); Aim 1a (PK study group 3); Aim 1a (PK study group 4); Aim 2a (Hybrid trial intervention group)
Drug: Etonogestrel (ETG) implant — Contraceptive progestin implants are thin rods inserted under the skin of a woman's arm
  Arms: Aim 1a (PK study group 2)
Drug: Intramuscular depo-medroxyprogesterone acetate (IM DMPA) — DMPA (150 mg of depo-medroxyprogesterone acetate (MPA)/ml IMI) is the most commonly used injectable contraceptive worldwide
  Arms: Aim 1a (PK study group 1); Aim 1a (PK study group 5)
Drug: Levonorgestrel — Contraceptive estrogen implants are thin rods inserted under the skin of a woman's arm
  Arms: Aim 1a (PK study group 3)
Drug: NNRTI, PI, or INSTI-containing 1st or 2nd line ART regimens — ART that concurrently contains combinations of non-nucleoside reverse transcriptase inhibitors (NNRTIs), such as efavirenz, and protease-inhibitors (PIs), such as atazanavir/ritonavir or lopinavir/ritonavir, or integrase inhibitors (INSTIs), such as raltegravir or dolutegravir
  Arms: Aim 2a (Hybrid trial comparator group)

SUMMARY:
The study investigators are conducting foundational pharmacokinetic (PK) and qualitative studies, among 15-24 years old (inclusive) adolescent girls and young women living with HIV (AGYWLHIV) already on oral antiretroviral therapy (ART) and virally suppressed, leading up to a hybrid type I effectiveness-implementation trial randomizing individual AGYWLHIV to receive long-acting (LA) injectable cabotegravir/rilpivirine vs. standard of care within one of Kenya's largest HIV treatment programs. The PK and qualitative studies will investigate potential issues arising from co-delivery and guide delivery of the effectiveness-implementation trial. The PK and qualitative studies will largely be conducted with a sentinel cohort of AGYWLHIV. Learning from this early LA ART use, the investigators will refine the procedures in the LA ART hybrid trial.

DETAILED DESCRIPTION:
Long-acting (LA) antiretroviral therapy (ART), such as injectable cabotegravir and rilpivirine, has been receiving global clinical approvals and has the potential to address barriers to ART and improve patient adherence and persistence to treatment. LA ART regimens can potentially also increase options for patients and providers to individualize treatment plans, provide a powerful treatment option for those experiencing adherence issues related oral treatment options, and may ease the burden of health systems in RLS. Another major threat to AGYW's health is unintended pregnancies and AGYWLHIV also face unique challenges in uptake and continuation of LA contraceptives. Use of LA ART may foster synergy in usage of LA contraceptives among AGYWLHIV.

This proposed research study has three main components: 1) a prospective, non-randomized, parallel-group pharmacokinetic (PK) study among a sentinel cohort of five distinct groups of AGYW, and will leverage existing control groups (Aim 1a); 2) a qualitative study that will conduct individual interviews with four different subgroups of AGYWLHIV from the sentinel cohort from the PK study, as well as focus group discussions with providers, policy makers, and other stakeholders for health systems readiness for wider scale-up (Aim 1b); and 3) an open-label, mixed methods, 48-week type I hybrid trial randomizing AGYW with viral suppression on their current ART regimen to switch to 1:1 cabotegravir/ rilpivirine (intervention arm) vs. continue their oral ART regimen (Aim 2a), with a component also evaluating implementation outcomes of acceptability, feasibility, and fidelity (Aim 2b). The proposed study will be conducted in HIV treatment facilities in western Kenya within the regional Moi Teaching and Referral Hospital (MTRH).

This study will provide foundational data for future studies and implementation plans related to addressing barriers and will critically inform follow-up studies of LA ART in other priority subpopulations. Providing an array of method options for both HIV treatment and pregnancy prevention has the potential to revolutionize personal decision-making and improve long-term outcomes for AGYWLHIV. Our real-world experiences of co-delivery will also inform future considerations for co-formulations of antiretrovirals and contraceptives for both HIV treatment and prevention.

Our central hypothesis is the following: 1) at the client level, the use of LA ART or contraceptives will foster long-term thinking for health, forging a convergence of the use of the two when applicable; and 2) at the program/provider level, leveraging existing LA contraceptive delivery platform will make LA ART highly acceptable, feasible, and deliverable with high fidelity.

Our overall objective in this study is to conduct the foundational PK and qualitative studies first as a lead in to the hybrid trial. Guided by Proctor et al.'s implementation outcomes framework, the hybrid trial will also focus on acceptability, feasibility, and fidelity. These implementation outcomes are proximal indicators of implementation processes and intermediate outcomes, which ultimately predict implementation success. Demonstrating successful implementation outcomes will then inform wider-scale implementation of LA ART, when service and client outcomes can be fully realized.

The PK and qualitative studies will investigate potential issues arising from co-delivery and guide delivery of the effectiveness-implementation trial. The PK (Aim 1a) and qualitative (Aim 1b) studies will largely be conducted with a sentinel cohort of AGYWLHIV in parallel to each other. Learning from this early LA ART use, the investigators will refine our procedures in the LA ART hybrid trial (Aim 2). For all possible outcomes/scenarios of Aim 1, the investigators still anticipate conducting a robust trial in Aim 2.

Thus, our specific aims are:

Aim 1: To collect foundational data to better inform design of an effectiveness-implementation trial.

Aim 1a: To determine if combined cabotegravir/rilpivirine injectable use has bidirectional drug-drug interactions with injectable (depot medroxyprogesterone acetate [DMPA]) or implantable (etonogestrel or levonorgestrel) contraceptives.

Aim 1b: To qualitatively explore points of convergence and divergence, preferences and values, and health systems readiness around wider-scale co-delivery of LA ART and contraceptives.

Aim 2: To evaluate the impact of clinic-provided, co-delivery of LA ART and contraceptives among AGYWLHIV.

Aim 2a: To evaluate the impact on effectiveness outcomes of HIV treatment (viral suppression and adherence/persistence) and contraception (uptake and continuation rates).

Aim 2b: To evaluate the impact on implementation outcomes of acceptability, feasibility, and fidelity.

ELIGIBILITY:
Inclusion Criteria (PK study):

* Female sex,
* HIV-positive (for PK groups #1-4) or HIV-uninfected (for PK group #5 only),
* Age 15-24 years at the time of enrollment,
* Documented or confirmed viral suppression for HIV (defined as <40 copies/mL) within 6 months prior to study enrollment,
* Have been on the study oral drug for at least 4 weeks for the PK groups #1-4,
* Have initiated and intends to use DMPA or implant for at least another three or 6 months, respectively,
* Willing to undergo phlebotomy every 4-12 weeks for the duration of the study period
* Able to consent or assent (with parental consent) for study participation in English or Kiswahili

Exclusion Criteria (PK study):

* Already be on ART that concurrently contains combinations of non-nucleoside reverse transcriptase inhibitors (NNRTIs), such as efavirenz, and protease-inhibitors (PIs), such as atazanavir/ritonavir or lopinavir/ritonavir, or integrase inhibitors (INSTIs), such as raltegravir or dolutegravir
* Currently pregnant or intends to become pregnant or breastfeeding within the next 12 or 24 weeks for DMPA or implant groups, respectively,
* Have had unprotected sex in the last two weeks or be currently pregnant via urine pregnancy testing,
* Use or anticipated use of drugs for the duration of the study period known to interact with hormonal implants or the study ART regimen,
* Current or planned concomitant use of other hormonal contraceptives,
* Be obese (BMI≥30),
* Evidence of Hepatitis B virus (HBV) infection based on the results of testing for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (anti-HBc), Hepatitis B surface antibody (anti-HBs) and HBV Deoxyribonucleic acid (DNA) as follows: positive for HBsAg being excluded or negative for anti-HBs but positive for anti-HBc (negative HBsAg status) and positive for HBV DNA are excluded (of note, participants positive for anti-HBc (negative HBsAg status) and positive for anti-HBs (past and/or current evidence) are immune to HBV and are not excluded).
* Serum ALT>5x ULN at the time of screening,
* Serum creatinine >2.5x ULN at the time of screening.

Inclusion Criteria Aim 1b (qualitative PK study):

* Participating in PK study for study participants,
* Self-identifying as provider, program person, policy-maker, or stakeholder relevant to the study topics, and age 18 years of age or older,
* Able to consent for study participation in English or Kiswahili

Inclusion Criteria (Hybrid trial):

* Female sex,
* HIV-positive,
* Age 15-24 years at the time of enrollment,
* Documented or confirmed viral suppression for HIV (defined as <40 copies/mL) within 6 months prior to study enrollment,
* Willing to undergo phlebotomy every 4-12 weeks for the duration of the study period,
* Able to consent or assent (with parental consent) for study participation in English or Kiswahili

Exclusion Criteria (Hybrid trial):

* Already be on ART that concurrently contains combinations of non-nucleoside reverse transcriptase inhibitors (NNRTIs), such as efavirenz, and protease-inhibitors (PIs), such as atazanavir/ritonavir or lopinavir/ritonavir, or integrase inhibitors (INSTIs), such as raltegravir or dolutegravir
* Currently pregnant or intends to become pregnant or breastfeeding within the next one year,
* Have had unprotected sex in the last two weeks or be currently pregnant via urine pregnancy testing,
* Use or anticipated use of drugs for the duration of the study period known to interact with the study ART regimen,
* Evidence of Hepatitis B virus (HBV) infection based on the results of testing for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (anti-HBc), Hepatitis B surface antibody (anti-HBs) and HBV Deoxyribonucleic acid (DNA) as follows: positive for HBsAg being excluded or negative for anti-HBs but positive for anti-HBc (negative HBsAg status) and positive for HBV DNA are excluded (of note, participants positive for anti-HBc (negative HBsAg status) and positive for anti-HBs (past and/or current evidence) are immune to HBV and are not excluded).
* Serum ALT>5x ULN at the time of screening,
* Serum creatinine >2.5x ULN at the time of screening.

Inclusion Criteria Aim 2b (qualitative study):

* Participating in hybrid trial study for study participants,
* Self-identifying as provider, program person, policy-maker, or stakeholder relevant to the study topics, and age 18 years of age or older,
* Able to consent for study participation in English or Kiswahili

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 700 (Estimated)
Dates: Start 2021-11-26 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Hormone concentrations with cabotegravir/rilpivirine use (Aim 1a) | 12 or 24 weeks after DMPA or implant initiation, respectively
  To assess differences in hormone concentrations with cabotegravir/rilpivirine use, the investigators will first calculate the progestin geometric mean concentrations at 12 or 24 weeks after DMPA or implant initiation, respectively, for each group. These geometric means will be compared to HIV-negative groups recruited in this study (for the DMPA comparator) or from the PARVI study (for the implants comparator), using geometric mean ratios with 90% confidence intervals (a FDA standard) and the Wilcoxon rank sum test.
Number of participants with HIV viral suppression (Aim 2a) | 48 weeks after study enrollment
  Our primary analysis will compare the proportion of participants with viral suppression (via HIV viral load <40 copies/mL) 48 weeks after study enrollment (primary outcome) in the intervention vs. control arms (primary exposure) using logistic regression, adjusting for age group strata.

SECONDARY OUTCOMES:
Adherence to ART (Aim 2a) | 3, 6, and 12 months after method initiation
  For secondary outcome of adherence to ART, the investigators will use multivariate logistic regression to assess associations between study arm and adherence/ medication possession ratio (MPR=[# pills dispensed - # pills returned]/[avg. # doses required per day * # days of use]) ≥95% over the preceding month prior to the VL evaluation.
Persistence to ART (Aim 2a) | 3, 6, and 12 months after method initiation
  For secondary outcome of persistence to ART, the investigators will use multivariate logistic regression to assess associations between study arm persistence/average MPR since study enrollment.
Contraceptive outcome (Aim 2a) | 3, 6, and 12 months after method initiation
  Among participants who are not already using a LA contraceptive method at enrollment and wish to delay pregnancy, the investigators will use Cox proportional hazards models to compare time to LA contraceptive uptake, or incident use, between study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Rena Patel, MD, MPH, MPhil, Principal Investigator — University of Alabama at Birmingham; Edwin Were, Principal Investigator — Moi Teaching and Referral Hospital; Edith Apondi, Principal Investigator — MTRH Adolescent Rafiki Clinic and Pediatric Program at AMPATH
Locations (1):
- Academic Model Providing Access to Healthcare (AMPATH) Moi Teaching And Referral Hospital (MTRH), Eldoret, Kenya, Kenya

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD that underlies the results reported in a publication will be provided. Data sharing will begin 9 months after article publication and will be available for up to 36 months. Data will be made available to qualified researchers whose proposed research has received IRB approval. The data will be provided through a data repository following the execution of a data-sharing agreement.
Supporting Information: Study Protocol
Time Frame: Starting 9 months and ending 36 months after article publication
Access Criteria: Investigators whose proposed use of the data has been approved by the investigators